CLINICAL TRIAL: NCT01628419
Title: Health Promotion Intervention Program at the Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: WIN12345
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Conditions Influencing Health Status
Keywords: Health promotion; Intervention; Workplace; Exercise program
MeSH Terms: interventions — Play Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health intervention program (Experimental): Health promotion intervention program will be implemented at each workplace and will include: exercise program, nutritional counseling for the kitchen service, lectures on different topics (physical activity, nutrition, sleeping behaviour etc.).
  Interventions: Behavioral: Health intervention

INTERVENTIONS:
Behavioral: Health intervention — physical activity program at the workplace - once a week with a certified trainer. (The program will include: aerobic exercises as well as resistance exercises). The employees will encourage to perform two additional workouts during the week.
  Nutritional counseling for the kitchen staff Lectures - lectures will be given at each worksite on different topics: physical activity, nutrition, sleeping behaviour, mental aspects.

SUMMARY:
The purpose of the current investigation is to examine the effects of health intervention program at the workplace on health risks for cardiovascular disease, well-being and absenteeism at the workplace.

Participants: 1500 male and female employees from 10 different companies across Israel will take part in the study. Age: older than 18 yrs.

Hypothesis 1: The intervention program will have positive effects on the health risks for cardiovascular disease. For example: Will be reflected in a decrease in LDL and increase in HDL.

Hypothesis 2: The intervention program will have positive effects on the absenteeism at the workplace (e.g. decrease in days of sick leave per employee).

DETAILED DESCRIPTION:
Introduction: The incidence of cardiovascular disease and related illnesses has been on the rise throughout the past decades. This increase is highly linked to a diet that is both high in calories and saturated fats as well as low levels of physical activity that may cause to an increase of body weight, percent of body fat and in some cases to obesity. It has been known that low levels of physical activity or sedentary behavior is a dominant risk factor for developing cardiovascular diseases.

At the work place, employees' work capacity and efficiency can highly be affected by a sedentary lifestyle and overweight conditions. A lack of physical activity was found to be associated with low levels of production at the workplace. Furthermore, a positive correlation was found between employees' lifestyle and number of days on a sick leave. Studies have shown that obesity and a lack of physical activity are significant risk factors for absenteeism.

In the past years, several studies have examined the effect of intervention programs on lifestyle behavior changes and the risk of developing cardiovascular diseases(CAD). The results of those studies are quite equivocal. Some have demonstrated a positive effect of the intervention programs on decreasing CAD risk factors and obesity rates, while others have found no clear effect. The conflicting results could be due to methodological issues and different studies' designs. For example, some studies did not report the amount and the intensity of the physical activity program used in the intervention program. Furthermore, some intervention programs did not include a nutritional manipulation. In a recent review papers, it was found that the most efficient programs were those that combined group workshops, guided physical activity programs and individualized counseling sessions for employers that were at a higher risk for developing CAD. Intervention program that included mainly guided physical activity were found to be less effective. It should be noted that the optimal program format that should be implemented at the workplace is not completely clear.

Study purpose: To examine the effect of health promotion intervention program at the workplace on risk factors to cardiovascular and metabolic diseases, well-being, life-style behavior and absenteeism at the workplace.

Subjects: The study will be approved by the local ethics committee. All participants will sign an informed consent form. Study's participants will include adult male and female (older than 18yrs). The 1500 participants will be recruited from 10 different worksites across Israel.

Study protocol: The length of the intervention program at each workplace will be 6 months. Parameters will be taken on two occasions: 1. Prior to the intervention program initiation 2. After 6 months.

Each employee at each workplace will be asked to fill a questionnaire regarding their medical history, life-style behavior, medications, physical activity habits, and nutrition and sleeping behavior. The employees will undergo anthropometric measurements and will be asked to perform blood test at Health maintenance organization (HMO). The same tests will perform at the end of the intervention program (after 6 months).

Anthropometric measures: subjects will be asked to wear light clothes. Height and weight will be measured with no shoes. Body Mass Index (BMI) will be calculated using the common formula (kg/m2). Circumference will be measured at two sites while the subject standing still with both feet close together. Waist circumference will be measured at the height of the bell-button; hip circumference will be measured at the widest point of the pelvis. Waist-hip ratio will calculate and compared to common and updated norms. Blood pressure and resting pulse will be measure twice while the subject is in a sitting position. The average value will be calculated.

Blood tests: Each participant in the study will be asked to perform the following tests prior to the beginning of the intervention program. The parameters will include: blood glucose, hemoglobin, LDL, HDL, cholesterol, triglycerides, liver function (GGT, ALT), Hemoglobin A1C.

Absenteeism from work (due to illnesses): With the assistance of the human resources department, at the end of the 6 months intervention program the number of days of sick leave will be recorded for each participant in the study. If applicable, data will be compared with last year absenteeism.

Intervention program characteristics: Structured and guided physical activity program with a certified trainer, General Guidelines for performing physical activity outside of working hours, Counseling and guidelines for the kitchen staff (in organization that has food services), Supplying general guidelines for healthy diet and nutrition, Modifying the working environment to a health promoting one (using posters, electronic communication, daily and weekly tips etc…), Lectures on general topics - physical activity, nutrition, ergonomics, behavior changes, sleeping behavior.

Structured physical activity program: The training program will include, a structured aerobic and resistance training session performed once a week with a certified trainer. The aerobic session will include running/walking for 20min in a moderate-vigorous intensity based on rate of perceived exertion scale from 1 (very light exercise) until 10 (very hard and strenuous exercise). During the first two weeks the intensity will remain relatively moderate (rate of perceived exertion 3-4), during the third week of the program the intensity will increase to 5-6 and from the fifth week on, the intensity will increase from 6 to 8.

The resistance training will include exercise for the major muscle groups for about 15-20 min. The resistance exercises will be performed with dumbbells, resistance bands and body weight. Additionally, the participants in the program will be asked to perform an additional aerobic workouts for 20-30min (rate of perceived exertion 5-6) during the week, at least two more workouts.

General guidelines for physical activity: All the participants in the study will receive pedometers for their personal use. All employees will receive the recommended amount of physical activity they should perform throughout the week. The information will be distributed through information sheets, posters and e-mails. The recommendations will include the different types of exercises that can be performed in order to improve aerobic fitness and the recommended doses such as: amounts of daily steps, amount of weekly steps. Furthermore, recommendations on strength, flexibility and core exercises will be provided.

Nutrition: In organizations that have food services and catering, certified dietitians from the Wingate Institute will advise the kitchen staff about healthy nutritional choices. Consultation will be given on the types of food to be served during meetings and events.

The professional staff will make sure that the organization provided equipment and means for employees to bring food from home, such as: refrigerators, microwaves or oven to warm up food, dining hall and cold water fountains.

A personal meeting will be available to the study's participants. In those meetings they will be able to discuss personal issues and received a personal diet plan.

General nutrition guidelines: General nutritional guidelines at the workplace and during free time will be provided to all employees. The information will be distributed through booklets, poster, information sheet and e-mails. The guidelines will include recommendation regarding healthy food choices, nutritional values of variety of food products, recommended recipes etc…

Promoting health at the workplace (modifying the working environment): A representative from the study group and the organization's management will map the working environment and will recommend possible modifications that can be performed to the working environment in order to make it a health promoting one. For example: improving the accessibility to spaces within the working environment where employees can exercise, informative signage and posters regarding healthy life-style choices, informative e-mails with weekly and monthly tips will send to the employees.

Lectures: As part of the intervention program the employees will receive 6 lectures dealing with different aspects of practicing a healthy life-style. The lectures will given by the professional staff from the Wingate Institute on difference topics, such as: healthy nutritional choices, ergonomics at the workplace, importance of performing physical activity, sleeping habits and working capacity, behavioral tools to make a life-style changes.

Statistical analyses: Paired t-test will be used to examine the intervention program effect on anthropometric measures, blood tests parameters and absenteeism. The effect of the intervention program will also be examined using multiple regressions analyses. Significant level will set at P<0.05. SPSS software will be used for all statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate in the study,
* older than 18 yrs

Exclusion Criteria:

* Missing blood tests results and anthropometric measures prior to the beginning of the study,
* unstable cardiac disease,
* unstable hypertension during rest (above 200 mmHg systolic blood pressure and above 110 mmHg of diastolic blood pressure),
* pregnancy,
* using pacemaker,
* past cardiac incidence during the 6 months preceding the test,
* other disease that might cause contraindication for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Anthropometric measures | 6 months
  The following measures will be evaluated: Height and body mass (Kg) and Body mass index will be calculated (BMI), hip and waist circumference and the ratio between the two measures will be calculated.

SECONDARY OUTCOMES:
Absenteeism from work | 6 months
  Number days of sick leave each employee had during the 6 months period.
Blood tests results | 6 months
  Improvement in Blood test results: blood glucose levels and Hemuglubin A1c, Hemoglubin, lipid profile (LDL, HDL, cholestrol, Triglycerides), liver function (ALT, GGT)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shargal, PhD, Study Director — Wingate Institute, Israel
Locations (1):
- Wingate Institute, Netanya, Israel